CLINICAL TRIAL: NCT06268795
Title: A Diagnostic Test Accuracy Study Comparing Biopsy to Aspiration in Shoulder and Elbow Arthroplasty Revision Surgery (BASE Study)
Status: Recruiting | Type: Observational
Sponsor: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: BASE
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Periprosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to compare the diagnostic accuracy of percutaneous aspiration against open biopsy, using microbiological and histological methods, for the detection of shoulder and elbow periprosthetic joint infection (PJI). This is to establish the utility of pre-operative joint aspiration in the treatment pathway for shoulder and elbow PJI.

DETAILED DESCRIPTION:
A PJI is a severe complication of arthroplasty surgery and one of the leading causes of revising joint replacements. It accounts for 19% of shoulder arthroplasty and 28% of elbow arthroplasty revisions. The successful management of patients with PJI depends on an early and accurate diagnosis, however, this can be challenging. To optimise the diagnosis of PJI, a combination of clinical findings, laboratory results from peripheral blood and synovial fluid (WBC and CRP), microbiological data, histological evaluation of periprosthetic tissue, intraoperative inspection, and radiographic results are considered.

Percutaneous joint aspiration makes an integral part of each of the diagnostic criteria for PJI (EBJIS, MSIS, ICM, and IDSA) and the current shoulder and elbow PJI guidelines from the British Elbow and Shoulder Society (BESS) state that a joint aspiration should be attempted in all patients. Aspiration allows for the identification of bacteria, the determination of antibiotic resistance and sensitivity patterns to guide anti-microbial management before surgery at relatively low costs, however, aspiration has a large variance in its diagnostic value. Studies have been performed to assess the diagnostic accuracy of percutaneous joint aspiration of suspected PJI in hip and knee arthroplasty but there is currently no evidence of utility in the diagnosis of PJI in shoulder and elbow arthroplasty.

The organisms causing PJI in shoulder and elbow arthroplasty may be different from lower limb arthroplasty and this may impact the accuracy of investigation findings. Cutibacterium (Propionibacterium) acnes is commonly isolated following upper limb surgery and is skin commensal. Therefore, distinguishing its presence as a pathogen can prove challenging due to its low virulence, limited local inflammatory response, biofilm formation, difficulty in culturing the bacteria and rising resistance rate to anti-microbial agents. This makes it even more essential that diagnostic tests can accurately identify causative PJI pathogens.

The gold standard for the diagnosis of PJI is open biopsy. This is usually performed by obtaining tissue samples intraoperatively. Radiologically guided biopsy is also recommended to be performed in certain cases e.g. not clinically confirmed PJI and surgery not feasible. To improve the diagnostic accuracy in suspected PJI of the shoulder and elbow, it has been hypothesised that pre-revision tissue biopsies, much like that for hip and knee arthroplasties, for microbiological and histological analyses are of superior diagnostic value than percutaneous aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 18 years or older.
* A participant is willing and able to give informed consent for participation in the study.
* Patient undergoing revision shoulder or elbow arthroplasty surgery.
* Previous anatomic total shoulder arthroplasty (TSA), shoulder hemiarthroplasty (HA), reverse total shoulder arthroplasty (RTSA), total elbow arthroplasty (TEA), distal humeral hemiarthroplasty (DHH) and radial head arthroplasty (RHA).

Exclusion Criteria:

* Refusal of consent.
* Antibiotic treatment was not stopped 2 weeks before aspiration or biopsy.
* Pregnancy.
* Part of any other trial with similar interventions unless previously agreed on with investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are 18 years or older that have been referred for potential revisions of the shoulder and elbow arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of diagnostic accuracy | 36 months
  Compare the diagnostic accuracy of percutaneous aspiration against the gold standard of open biopsy with multiple tissue samples

SECONDARY OUTCOMES:
Culture analysis | 14 days
  To determine the sensitivity, specificity, positive/negative predictive value, negative, diagnostic accuracy & positive/negative likelihood ratios of needle aspiration and open biopsy for the diagnosis of periprosthetic joint infection in shoulder and elbow replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Wrightington Wigan & Leigh Teaching Hospitals NHS Foundation Trust, Wigan, Lancashire, United Kingdom